CLINICAL TRIAL: NCT06425107
Title: Point-of-Care Lung Ultrasound for Prognosis in Critically Ill Infants With Acute Lower Respiratory Tract Infection
Acronym: Bacon-Pocus
Status: Recruiting | Type: Observational
Sponsor: Vittore Buzzi Children's Hospital (Other)
Responsible Party: Principal Investigator, Anna Camporesi, Principal Investigator, Vittore Buzzi Children's Hospital
Other Study IDs: CET 23-2024
Record Dates: First submitted 2024-05-09; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Bronchiolitis; Noninvasive Ventilation
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective, observational multicentric study which aims at identifying lung POCUS (Point of Care UltraSound) findings associated with failure of noninvasive ICU-LRS (Intensive Care Unit Level Respiratory Support) (defined as escalation of settings or need for intubation and invasive mechanical ventilation) in infants requiring noninvasive ICU-LRS in the ICU for bronchiolitis and other LRTI (Low Respiratory Tract Infection) and at identifying lung, pleural, and diaphragm POCUS findings that are associated with a clinical improvement after escalation of ICU-LRS support by comparing POCUS findings from the first 24 hours of ICU stay to a subsequent study 1 day later.

DETAILED DESCRIPTION:
Lower respiratory tract infections, primarily viral bronchiolitis, are a common cause of PICU admission for infants. While overall hospitalization rates for bronchiolitis are declining, ICU admission rates are actually increasing. The trend in respiratory management of critically ill infants with LRTIs has shifted from frequent invasive mechanical ventilation to more common use of non-invasive modalities, including CPAP, BiPap, and HFNC. Currently, the overwhelming majority of infants requiring ICU-level respiratory support (ICU-LRS) for bronchiolitis receive only noninvasive support.

During the past decade, point-of-care lung ultrasound (POCUS) is increasingly being used in both adults and children to enhance diagnostic and prognostic ability in respiratory failure. Lung POCUS is appealing due to the lack of radiation exposure compared to x-rays, the added sensitivity and specificity that it can add compared to traditional imaging to help differentiate consolidation from atelectasis from edema (may all have similar appearance on x-rays), the dynamic nature of the study to evaluate the lung parenchyma, pleura, and diaphragm, and the fact that it can be easily applied and repeated at the bedside to guide adjustments to therapies and evaluate their response. Lung POCUS differs from traditional radiology-based lung ultrasound in that it is focused and goal-directed, is frequently performed serially by the clinician managing the patient at the bedside, and is frequently used to immediately direct care decisions in real-time.

While lung POCUS is quickly becoming a standard of care for adults with respiratory failure, pediatric data, particularly in critically ill infants with bronchiolitis and other lower respiratory tract infections (LRTI) is largely lacking. Investigators from some sites within the BACON research group have begun to evaluate the role of lung POCUS in infants with bronchiolitis. These studies have primarily focused on the emergency department, but they have identified POCUS findings that are associated with clinical deterioration and have developed a pediatric lung ultrasound score that can predict infants who will require ICU-LRS. There are only two pediatric ICU bronchiolitis studies-one looking at the lung/pleura but in invasively ventilated patients only, and the other focused on the diaphragm in patients requiring noninvasive support.

Unfortunately, there are minimal data on infants in the ICU with bronchiolitis, and all of these prior studies are limited by low sample size. Thus, there is a significant knowledge gap about the ability of lung POCUS and these previously identified findings and scoring systems to accurately predict failure of noninvasive ICU-LRS for infants in the ICU with bronchiolitis and other LRTIs. Furthermore, there are no data evaluating the role of lung POCUS in identifying patients who will have a favorable response to adjustments in ICU-LRS settings.

Endpoints of the study are:

1, To identify lung POCUS findings associated with failure of noninvasive ICU-LRS (defined as escalation of settings or need for intubation and invasive mechanical ventilation) in infants requiring noninvasive ICU-LRS in the ICU for bronchiolitis and other LRTI.

2. To identify lung, pleural, and diaphragm POCUS findings that are associated with a clinical improvement after escalation of ICU-LRS support by comparing POCUS findings from the first 24 hours of ICU stay to a subsequent study 1 day later.

There are no specific safety endpoints for this observational study. Families could end participation by their infant at any time, and the treating physician or investigator could withdraw the patient from the study but there are no pre-specified safety endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Age <1 year at the time of hospital admission
2. Admission to PICU for suspected/confirmed LRTI
3. Treatment (within the 1st 12 hours of ICU stay) with noninvasive ICU-LRS for respiratory failure (HFNC >1L/kg/min, negative pressure, or noninvasive PPV via any interface (CPAP, BiPap, NIMV, etc.)

Exclusion Criteria:

1. Invasive ventilation as initial support or within the 1st 12 hours of ICU stay, either via endotracheal tube or tracheostomy
2. Upper respiratory symptoms only (stridor, stertor)
3. Corrected gestational age <37 weeks at time of ICU admission
4. ICU-LRS for only nonrespiratory reasons (e.g. shock) or for pulmonary edema felt to be solely due to noninfectious causes (cardiogenic, airway obstruction, drowning). Patients presenting with apnea can be included if they have a diagnosis of bronchiolitis or other LRTI
5. Prior inclusion in the study

Ages: 0 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants <1 year old admitted to the ICU for bronchiolitis and other lower respiratory tract infection who require noninvasive respiratory support
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Lung Ultrasound findings associated with failure of noninvasive ICU-LRS (defined as escalation of settings or need for intubation and invasive mechanical ventilation) in infants requiring noninvasive ICU-LRS in the ICU for bronchiolitis and other LRTI. | First 24 hours after ICU admission
  Ultrasound findings will be graded according to the scale proposed by the Italian Academy of thoracic Ultrasound: 0: normal A lines
  1. short vertical artifacts and isolated B lines
  2. multiple B lines (B lines with a distance of less than half centimeter to the confluence, remaining identifiable from each other)
  3. white lung (subpleural field with various shades of grey/white without distinguishing B lines) and subpleural consolidations smaller than 1 cm
  4. subpleural consolidations bigger than 1 cm

CONTACTS AND LOCATIONS:
Locations (1):
- Vittore Buzzi Children's Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caiulo VA, Gargani L, Caiulo S, Fisicaro A, Moramarco F, Latini G, Picano E. Lung ultrasound in bronchiolitis: comparison with chest X-ray. Eur J Pediatr. 2011 Nov;170(11):1427-33. doi: 10.1007/s00431-011-1461-2. Epub 2011 Apr 6. PMID 21468639
- [Background] Gori L, Amendolea A, Buonsenso D, Salvadori S, Supino MC, Musolino AM, Adamoli P, Coco AD, Trobia GL, Biagi C, Lucherini M, Leonardi A, Limoli G, Giampietri M, Sciacca TV, Morello R, Tursi F, Soldati G, Ecobron Group. Prognostic Role of Lung Ultrasound in Children with Bronchiolitis: Multicentric Prospective Study. J Clin Med. 2022 Jul 21;11(14):4233. doi: 10.3390/jcm11144233. PMID 35887997
- [Background] Musolino AM, Toma P, De Rose C, Pitaro E, Boccuzzi E, De Santis R, Morello R, Supino MC, Villani A, Valentini P, Buonsenso D. Ten Years of Pediatric Lung Ultrasound: A Narrative Review. Front Physiol. 2022 Jan 6;12:721951. doi: 10.3389/fphys.2021.721951. eCollection 2021. PMID 35069230
- [Background] Amendolea A, Gori L, Adamoli P, Limoli G, Supino MC, Coco AD, Trobia GL, Tursi F, Soldati G, Buonsenso D; Gruppo di studio Pediatrico AdET. Pleuropulmonary Ultrasound in Pediatrics: Proposal of a Reporting Model From the Academy of Thoracic Ultrasound. J Ultrasound Med. 2022 Oct;41(10):2637-2641. doi: 10.1002/jum.15924. Epub 2021 Dec 29. PMID 34964991